CLINICAL TRIAL: NCT00403598
Title: Preliminary Study for Identification of Calcium-Binding Proteins in the Serum in Various Metabolic Bone Disorders
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Ben-Gurion University of the Negev (Other)
Other Study IDs: SHEBA-06-4372-IV-CTIL
Record Dates: First submitted 2006-11-23; First posted 2006-11-27 (Estimated); Last update posted 2006-11-27 (Estimated); Status verified 2006-11

CONDITIONS: Osteoporosis; Osteitis Deformans; Parathyroid Diseases
MeSH Terms: conditions — Osteoporosis; Osteitis Deformans; Parathyroid Diseases

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
The purpose of this study is to determine whether the serum levels of certain calcium-binding proteins may be helpful in the diagnosis and management of metabolic bone diseases.

DETAILED DESCRIPTION:
Osteoporosis is an important and costly health issue. The diagnosis of the disease is based on measurement of bone mineral density or the occurrence of characteristic fractures. Currently it is not possible to predict fractures in individual patients, and the ability to monitor the response to treatment is limited as well.

We have synthesized and characterized a novel photoreactive Ca2+-analog reagent, Azido ruthenium (AzRu) that binds covalently to Ca2+-binding sites in proteins. The specificity of AzRu for Ca2+-binding proteins, its photoactivation and its radioactive labeling pave the way for a wide use of AzRu as a powerful tool to assess Ca2+-dependent cellular processes, both in vitro and in vivo. Using radiolabeled AzRu, it will be possible to identify Ca2+-binding proteins in a biological sample such as whole cell, isolated mitochondria, ER or other protein containing fractions. Protein bound [103Ru]AzRu in biological sample can be separated by SDS gel electrophoresis, followed by Coomassie staining and exposure of the dried gel to X-ray film (autoradiography). This allows the identification of the [103Ru] radiolabeled proteins. The labeled protein bands can be cut from the gel and subjected to MALADI-TOF analysis and the identity of the protein can be determined by a sequence homology search.

These would allow detection of Ca2+-binding proteins in the serum of various diseases and disorders, potentially leading to identification of novel biomarkers for disease diagnostics.

We would like to use blood samples to carry out the procedure described above for identification of Ca2+ binding proteins appearing or their level is increased in disease or under pathogenic conditions. Since Ca2+ binding proteins play an important role in bone metabolism, we chose to test their occurrence in the serum of patients with osteoporosis and other metabolic bone diseases.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of a metabolic bone disorder

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Iris Vered, M.D, Principal Investigator — Sheba Medical Center, Tel Hashomer
Locations (1):
- Sheba Medical Center, Tel Hashomer, Ramat Gan, Israel